CLINICAL TRIAL: NCT06374888
Title: A Single-arm, Open, Multicenter Phase II Clinical Study of Nilatinib Maleate Tablets Combined With Capecitabine in the Treatment of HER2-positive Advanced Esophageal/Esophagogastric Junction/Gastric Adenocarcinoma With Brain Metastases
Brief Title: Nilatinib Maleate Tablets Combined With Capecitabine in the Treatment of HER2-positive Advanced Esophageal/Esophagogastric Junction/Gastric Adenocarcinoma With Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL009-2002
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Her2-positive Advanced Esophageal/Esophagogastric Junction/Gastric Adenocarcinoma With Brain Metastasis
Keywords: Her2-positive; esophageal; esophagogastric junction; gastric adenocarcinoma; brain metastasis
MeSH Terms: conditions — Brain Neoplasms | interventions — neratinib; Capecitabine

STUDY DESIGN:
Intervention Model Description: Her2-positive advanced esophageal/esophagogastric junction/gastric adenocarcinoma with brain metastases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Cohort A: : Patients with brain metastases who had not previously received central nervous system radiotherapy, distance from the last systemic treatment junction The beam should be longer than 2 weeks. Cohort B: Patients with disease progression or new lesions after whole brain radiotherapy or stereotactic radiotherapy; For accepted offices For partially treated lesions, there is clear evidence of progress in imaging examination, and the lesions that have received radiotherapy can be selected as target diseases
  Interventions: Drug: Neratinib maleate in combination with capecitabine

INTERVENTIONS:
Drug: Neratinib maleate in combination with capecitabine — Neratinib maleate tablets，Tablets, 40mg/ tablet, 180 tablets/bottle, orally, 240mg once daily, sealed, stored not above 25℃

SUMMARY:
To evaluate the efficacy of nilatinib maleate tablets combined with capecitabine in the treatment of HER2-positive advanced esophageal/esophagogastric junction/gastric adenocarcinoma with brain metastasis.

DETAILED DESCRIPTION:
Twenty-eight patients with HER2-positive gastric cancer with brain metastasis were divided into two cohorts： Cohort A: Patients with brain metastases who have not previously received central nervous system radiotherapy, distance from the last systemic treatment junction The beam should be longer than 2 weeks. Cohort B: Patients with disease progression or new lesions after whole brain radiotherapy or stereotactic radiotherapy; For accepted offices For partially treated lesions, there is clear evidence of progress in imaging examination, and the lesions that have received radiotherapy can be selected as target diseases The kitchen range.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Histologically or cytologically confirmed advanced esophageal/esophagogastric junction/gastric adenocarcinoma with brain metastases (clear imaging evidence of metastasis)
* Tumor tissue was HER2 positive Her2-positive is defined as immunohistochemical (IHC) 3+ or IHC 2+ and in situhybridization (ISH) positive
* Presence of a measurable lesion according to RECIST 1.1: presence of at least one non-radiation-treated lesion with a diameter ≥10 mm (lymph node lesion with a diameter ≥15 mm) that can be accurately measured at baseline on CT or MRI and can be repeatedly measured. If study participants only have lesions after radiotherapy, and the lesions have been clearly identified as radiological progression and can be measured, they can be selected as target lesions. The brain lesion must have a measurable target lesion, but it is not required to have a measurable targetlesion outside the brain
* Corticosteroid dose did not increase one week before brain MRI examination
* There is no limit to previous treatment options, including chemotherapy, radiotherapy, targeted drugs, antibody coupling drugs, immunosuppressants, etc
* Cohort A: Patients with brain metastases who have not previously received central nervous system radiotherapy should be more than 2 weeks from the end of the last systemic therapy. Patients who developed new brain lesions after craniotomy were allowed to be included if they had not received postoperative radiotherapy and were at least 2 weeks removed from surgery.

Cohort B: Patients with disease progression or new lesions after whole brain radiotherapy or stereotactic radiotherapy; For lesions that have received local treatment, there is clear evidence of progress in imaging examination, and those that have received radiotherapy can be selected as target lesions. Patients with multiple central nervous system lesions, only one or a few of which received stereotactic radiotherapy, and those with lesions that did not receive local treatment, may still participate in the study

* Predicted survival ≥8 weeks
* Women of reproductive age should agree to use contraceptives (such as Iuds, contraceptives or condoms) during the study period and for 6 months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be a non-lactating patient; Men should consent to patients who must use contraception during the study period and for 6 months after the end of the study period
* The patient can understand the situation of this study, and the patient and (or) legal representative voluntarily agree to participate in this trial and sign the informed consent

Exclusion Criteria:

* Participants who have received chemotherapy or radiation therapy (including study drugs) within 2 weeks prior to study participation, or who have not fully recovered from adverse events (excluding hair loss) due to taking drugs for more than 4 weeks
* Patients who have previously received anti-HER2 small-molecule TKI therapy progression
* More than two seizures in the first 4 weeks of enrollment
* Participants currently receiving any other study drug
* History of allergic reactions caused by compounds chemically or biologically similar to neratinib
* Concurrent use of enzyme-induced antiepileptic drugs (EIED), including phenytoin, carbamazepine, oxamazepine, phophenytoin, phenobarbital, pentobarbital, or primidone
* Patients who were receiving any concurrent treatment for cancer during the study period, such as concurrent chemotherapy, radiation, or hormone therapy. Concurrent treatment with bisphosphonates is permitted, but should be started before the first dose of nelatinib
* Present with co-existing medical conditions, including but not limited to persistent or active infections, symptomatic congestive heart failure, unstable angina, arrhythmia, or mental illness/social conditions that would limit compliance with study requirements
* Patients with known contraindications to MRI, such as pacemakers, shrapnel, or ocular foreign bodies
* Patients with pial metastasis only
* Severe malabsorption syndrome or inability to tolerate oral drugs
* Any chronic disease that causes diarrhea with CTCAE≥2 at baseline
* Women who are breastfeeding or whose blood or urine pregnancy test results are positive within 7 days before the first dosing of the study treatment
* The investigators identified patients with any conditions that compromised patient safety, interfered with study evaluation, or had poor adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rates of the central nervous system as assessed by the Independent Imaging Evaluation Committee based on RECIST1.1 | Throughout the study for approximately 3.5 years
  Objective response rates: Proportion of patients whose tumor volume shrinks by 30% and is maintained for more than 4 weeks

SECONDARY OUTCOMES:
Central nervous response rate | Throughout the study for approximately 3.5 years
  reference to RANO-BM evaluation criteria for neurologic tumor brain metastases
Objective response rates outside the central nervous system | Throughout the study for approximately 3.5 years
  ORR,Proportion of patients with a 30% reduction in tumor volume that lasts more than 4 weeks
Disease control rate | Throughout the study for approximately 3.5 years
  It refers to the proportion of cases with complete response, partial response, and stable disease after treatment
Duration of reaction | Throughout the study for approximately 3.5 years
  It refers to the time between the first evaluation of a tumor as CR or PR and the second evaluation as Progressive Disease (PD) or death from any cause.
Clinical benefit rate | Throughout the study for approximately 3.5 years
  Refers to the time from the first evaluation of a tumor as CR or PR to the first evaluation as PD or death from any cause.
overall survival | Throughout the study for approximately 3.5 years
  Refers to the time between the start of treatment and the patient's death or last follow-up.

IPD SHARING:
Plan to Share IPD: No